CLINICAL TRIAL: NCT00280852
Title: A Retrospective Review of Multimodality Management of Anaplastic Thyroid Cancer
Brief Title: Review of Multimodality Management of Anaplastic Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Other Study IDs: 18940
Record Dates: First submitted 2006-01-20; First posted 2006-01-24 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-07

CONDITIONS: Anaplastic Thyroid Cancer
Keywords: anaplastic thyroid cancer; chemotherapy; radiotherapy
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
To describe the outcome of patients with anaplastic thyroid cancer treated with hyperfractionated radiotherapy and concomitant chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* anaplastic thyroid cancer treated with multimodality treatment

Exclusion Criteria:

* differentiated thyroid cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: anaplastic thyroid cancer
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2006-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold Lau, MD, Principal Investigator — Alberta Cancerboard
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada